CLINICAL TRIAL: NCT00648102
Title: A Phase I, Open-Label, Dose-Escalation, Multidose Study of CDX-1307, a Mannose Receptor-Targeted hCG-β Vaccine, in Patients With Incurable Locally Advanced or Metastatic Breast, Colorectal, Pancreatic, Bladder and Ovarian Cancer
Brief Title: Phase I Study of CDX-1307, hCG-B Vaccine, for Patients With Incurable, Locally Advanced or Metastatic Breast, Colorectal, Pancreatic, Bladder or Ovarian Cancer
Acronym: CDX1307-02
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: National Institute of Health, Celldex Therapeutics, Celldex Therapeutics
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDX1307-02
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Last update posted 2010-07-26 (Estimated); Status verified 2010-07

CONDITIONS: Breast Cancer; Colorectal Cancer; Pancreatic Cancer; Bladder Cancer; Ovarian Cancer
Keywords: Breast cancer; Colorectal cancer; Pancreatic cancer; Bladder cancer; Ovarian cancer; Metastatic cancer; Locally advanced cancer; Cancer Vaccine; Vaccine
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms; Urinary Bladder Neoplasms; Ovarian Neoplasms; Neoplasm Metastasis | interventions — CDX 1307

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: CDX-1307

SUMMARY:
This research study is for individuals who have advanced breast, colon, pancreatic, ovarian or bladder cancer. Celldex Therapeutics, Inc. is testing a form of immune therapy (vaccine) to see if it can be used to make the immune system attack the cancer. The study includes administration of additional treatments, in combination, thought to enhance the immune response effect. This study specifically administers the vaccine systemically to explore whether dendritic cell targeted vaccines can generate more robust effects via intravenous injection. (CDX 1307-02)

DETAILED DESCRIPTION:
Protocol CDX1307-02: CDX-1307 is an investigational drug that is being tested to see if it can stimulate the immune system (the cells and substances that protect the body from infection and foreign matter) of people with certain kinds of cancer. It is believed that the body's immune system can attack tumor cells and kill them. It is thought that immune cells recognize special proteins on the surface of tumors as a signal to fight the cancer. One of these proteins is called human chorionic gonadotropin-beta (hCG-β) and is found on several types of cancers including breast, colorectal, pancreatic, bladder and ovarian. The study drug, CDX-1307, is given as an intravenous infusion (administered in a vein in the arm or through a port-a-catheter). In addition, the study includes combination therapies which are thought to stimulate the immune response against tumor cells. In addition, the study includes combination therapies which are thought to stimulate the immune response against tumor cells.

ELIGIBILITY:
Inclusion Criteria

1. Patients must have incurable, metastatic or unresectable locally advanced breast, colorectal, pancreatic, bladder or ovarian cancer with measurable or evaluable-only disease. Locally advanced breast cancer is defined as inflammatory breast cancer with biopsy-proven skin involvement, or chest wall recurrence. Locally advanced disease of other histologies is defined according to the standard definition for that disease. Evaluable-only disease includes bone only or unresectable skin/chest wall only metastases, but does not include malignant effusion(s) only. Cancer with elevated serum tumor marker(s) (e.g. CA27.29, carcinoembryonic antigen, etc.) only does not constitute evaluable disease.
2. Patients must be 18 years of age or older.
3. Both genders may be enrolled.
4. At least 4 weeks must have elapsed between prior therapy and initiation of treatment with CDX-1307. Prior radiation therapy must be completed at least 4 weeks prior to enrollment. No prior radiopharmaceuticals within 8 weeks prior to enrollment. The patient must have recovered from any clinically significant toxicity experienced during prior treatment(s).
5. Patients on the following medications may be enrolled into the study if the medications were initiated ≥ 8 weeks prior to Screening and if no dosing changes are anticipated during the study:

   1. Hormonal therapy including gonadotropin releasing hormone (GnRh) agonist, antiandrogens, selective estrogen receptor modulators (SERMs), aromatase inhibitors, and progestins.
   2. Bisphosphonates.
6. Patients must have an ECOG Performance Status of 0 or 1.
7. Breast cancer patients must have received and progressed through at least one line of chemotherapy or endocrine therapy for metastatic or unresectable locally advanced breast cancer. Patients with HER2-positive breast cancer must have received and progressed through at least one line of chemotherapy plus trastuzumab, or endocrine therapy plus trastuzumab, for metastatic or unresectable locally advanced breast cancer. For incurable colorectal, pancreatic, bladder, or ovarian cancer, where therapy with potential survival benefit is available or where disease-specific palliation is the goal of therapy, patients must have received these appropriate standard of care therapies and experienced recurrence or progression while on that care. If no such therapy is available, patients with progressive disease may be enrolled. Chemotherapy or radiation must be discontinued at least 4 weeks prior to initiation of vaccination with CDX-1307.
8. Patients must have a life expectancy ≥ 16 weeks.
9. Male patients who are sexually active must agree to practice an effective form of barrier contraception during the course of the study.
10. Screening laboratory values must meet the following criteria:

    * Neutrophils ≥1.5 x109/L
    * Platelets >100 x109/L
    * Hemoglobin ≥10 g/dL
    * Creatinine <2 mg/dL
    * AST ≤2 X ULN
    * Bilirubin ≤2 X ULN unless due to Gilbert's syndrome.

      * Laboratory abnormalities attributed to liver involvement with cancer but outside of the normal range will be allowed if they do not exceed the following limits:
    * AST ≤4 X ULN

Exclusion Criteria

1. Since treatment with CDX-1307 theoretically may cause permanent sterility, women of childbearing potential will be excluded. Women who participate in this study must be post-menopausal [absence of menses for at least 2 years or age >55] and/or surgically incapable of bearing children.
2. Previous administration of hCG-β vaccine or therapy.
3. Concurrent treatment with immunosuppressive or immunomodulatory agents.
4. Positive tests for HIV, HBV or HCV.
5. Patients with systemic infection within 72 hours of registration that require antibiotics or produce a fever > 101oF.
6. Patients with active central nervous system metastases, unless previously treated and asymptomatic and not progressive in size or number for 2 months (1 month in the case of stereotactic radiation).
7. History of a second malignancy, except for adequately treated and cured basal or squamous cell skin cancer or cervical cancer in situ; or any other cancer from which the patient has been disease-free for ≥ 5 years.
8. History of anaphylactic reaction following exposure to humanized or human therapeutic monoclonal antibodies, or known hypersensitivity to GM-CSF or yeast derived products.
9. Patients with any of the following conditions: myocardial infarction within 1 year of Screening, congestive heart failure (unless LVEF ≥ 50% as determined by MUGA within 30 days of Screening), uncontrolled hypertension (≥ 160 mm Hg/systolic and ≥ 100 mm Hg/diastolic), symptomatic or life-threatening arrhythmia persistent on medication at Screening, or clinically evident chronic lung disease unless lung capacity ≥ 55% or FEV1 ≥ 60% at Screening. Note that the performance of MUGA scans and Pulmonary Function Tests are not required except if clinically indicated.
10. Any underlying medical condition that in the Principal Investigator's opinion will make the administration of study drug hazardous to the patient or would obscure the interpretation of adverse events.
11. Medical condition requiring the use of corticosteroids (must be discontinued at least 4 weeks prior to enrollment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2006-01; Primary Completion 2009-05 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To establish safety and tolerability profile of CDX1307 alone and with adjuvant in patients with breast, colorectal, pancreatic, bladder and ovarian cancer | up to 2 years or until progression

SECONDARY OUTCOMES:
Investigate clinical activity | up to 2 years or until progression

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Henry Ford Health System, Detroit, Michigan
  - Duke University, Durham, North Carolina
  - Carolina BioOncology Institute, Huntersville, North Carolina